CLINICAL TRIAL: NCT06996977
Title: The Effect of Menstrual Cycle on Postanesthetic Shivering; Prospective Observational Study
Brief Title: Menstrual Cycle and Postanesthetic Shivering
Status: Not yet recruiting | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Halide Hande Şahinkaya, Principal Investigator, Bozyaka Training and Research Hospital
Other Study IDs: menstrual cycle
Record Dates: First submitted 2025-05-07; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Shivering
Keywords: menstrual cycle; core temperature

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group follicular: Follicular phase of menstrual cycle
- Group luteal: Luteal phase of menstrual cycle

SUMMARY:
The goal of this observational study is to learn about the effect of menstrual cycle on postoperative shivering in women of fertile age. The main question it aims to answer is:

- Do women in the luteal phase have less postoperative shivering? Participants will have their intraoperative body temperature recorded and will be observed for postanesthetic shivering, depending on whether they are in the luteal phase or follicular phase.

DETAILED DESCRIPTION:
Postoperative shivering is a protective mechanism that the body uses to raise body temperature by rhythmic muscle contractions during hypothermia. Peroperative hypothermia is the most important cause of shivering after recovery. Shivering not only causes a decrease in patient comfort and discomfort but also increases metabolic demand by increasing oxygen consumption. This is an undesirable situation.

Women's hormonal status affects body temperature control. During the luteal phase, progesterone levels increase and this results in a 0.4 °C increase in core body temperature. The threshold for vasodilation also increases during this phase. Therefore, thermoregulation also changes during the luteal phase. Core body temperature in the follicular and luteal phase does not change with exposure to cold. However, under general anesthesia, core temperature is significantly reduced in both the luteal and follicular phase. Thermoregulatory vasoconstriction is less inhibited during luteal phase anesthesia.

The primary aim of our study was to determine the relationship between different phases of the menstrual cycle and the frequency of postoperative shivering. The secondary aim was to evaluate the incidence of intraoperative hypothermia and the duration of onset of intraoperative hypothermia in different phases of the menstrual cycle.

The study is planned as a prospective cross-sectional observational study. Female patients aged 18-45 years with ASA (American Society of Anesthesiology) score I-II who will undergo elective surgery for open technique septoplasty or rhinoplasty will be included in the study. They will be recorded in two groups as follicular group (F) and luteal group (L).

Patients data will be recorded;

* Demographic data
* Primary disease
* Comorbidities
* American Society of Anesthesiologists (ASA) Physical Status Classification
* The phase of the menstrual cycle (luteal or follicular phase) according to the patient's medical history
* Core body temperatures will be noted in the preoperative waiting area, before induction of general anesthesia, 1st hour under general anesthesia, 2nd hour under general anesthesia, 3rd hour under general anesthesia and in the postanesthetic recovery unit.
* Anesthesia and duration of surgery
* Infusion fluid quantity
* Pain level in the postoperative recovery unit (numerical rating scale-NRS)
* Postoperative tremors
* PAS (postanesthetic shivering scale) value SPSS statistical program for Windows will be used for statistical analysis of the results. Considering the number of surgeries performed in previous periods, it was predicted that approximately 100 patients could be included in the study within this period. This period, which was determined to ensure homogeneous distribution of the groups, will be extended if necessary and more patients will be included in the study. Parametric descriptive values will be given as mean and standard deviation, and non-parametric values will be given as n (%) and median and IQR (interquartile range). The conformity of the data to normal distribution will be evaluated by one sample Kolmogorov-Smirnov test. Comparisons of quantitative data conforming to normal distribution will be made with Student T test and comparisons of data not conforming to normal distribution will be made with Mann Whitney U test. Chi-Square test will be used to compare qualitative data. For the analyses, the significance level will be accepted as p<0.05 at 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Female patients undergoing elective open technical septoplasty or rhinoplasty
* 18-45 years of age
* ASA score I-II

Exclusion Criteria:

* Patient-legal representative does not want to be included in the study
* Emergency surgery
* Use of drugs that affect cardiovascular function, heat balance and hormone levels (e.g. combined oral contraceptives)
* Menstrual irregularity
* Polycystic ovary syndrome
* Thyroid disease
* Autonomic disease
* Reyno disease
* Uncontrolled diabetes mellitus
* Uncontrolled hypertension
* Surgeries where the duration of anesthesia is less than 1 hour
* Patients with NRS pain score above 7 in the recovery unit after anesthesia
* Core body temperature below 36°C before induction of general anesthesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patients scheduled for elective nose surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative Shivering | First 15 minutes after surgery
  Postanesthetic shivering will be evaluated in the postanesthesia care unit by Postanesthetic Shivering Scale. The scale is a 5-points scale. 0= no shivering
  1= no visible muscle activity but piloerection, peripheral vasoconstriction, or both are present (other causes excluded); 2 = muscular activity in only one muscle group; 3 = moderate muscular activity in more than one muscle group but no generalized shaking; 4 = violent muscular activity that involves the whole body. 3 and 4 mean worse outcome as the patient needs medication to treat shivering.
Number of patients who require meperidine | first 15 minutes after surgery
  The need for intravenous meperidine administration when the postanesthetic shivering scale (PAS) of the patient is above 3.

SECONDARY OUTCOMES:
Number of patients whose core body temperature is below 36 °C | perioperative
  Intraoperative hypothermia is defined as a core body temperature below 36°C under anesthesia.
The time when intraoperative core body temperature is detected below 36 °C | perioperative
  The time when the core body temperature is below 36°C during general anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Halide Hande ŞAHİNKAYA, MD, Principal Investigator — Izmir City Hospital; Gözde GÜRSOY ÇİRKİNOĞLU, MD, Study Chair — Izmir City Hospital; Tuba KUVVET YOLDAŞ, MD, Study Chair — Izmir City Hospital; Volkan HANCI, MD, Study Chair — 9 Eylul University Faculty of Medicine
Locations (1):
- Izmir City Hospital, Izmir, Bayraklı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Simegn GD, Bayable SD, Fetene MB. Prevention and management of perioperative hypothermia in adult elective surgical patients: A systematic review. Ann Med Surg (Lond). 2021 Nov 14;72:103059. doi: 10.1016/j.amsu.2021.103059. eCollection 2021 Dec. PMID 34840773
- [Background] Tatsumi T, Sampei M, Saito K, Honda Y, Okazaki Y, Arata N, Narumi K, Morisaki N, Ishikawa T, Narumi S. Age-Dependent and Seasonal Changes in Menstrual Cycle Length and Body Temperature Based on Big Data. Obstet Gynecol. 2020 Oct;136(4):666-674. doi: 10.1097/AOG.0000000000003910. PMID 32925608
- [Background] 1. V. Erden, C. Güler, H. Bulut, N. Özsoy Toprak, and N. Uslu, "Menstrual cycle phase may effect the thermoregulation during anesthesia," International Journal of Anesthesia, vol. 5, 2018.